CLINICAL TRIAL: NCT06403137
Title: The Effectiveness of Daily Protein Supplementation With a Plant Protein Blend or Milk Protein to Support Integrated Muscle Protein Synthesis Rates With and Without Exercise in Healthy Older Individuals
Brief Title: Plant Protein Blend and Milk Protein Supplements in Older Individuals
Acronym: Blend-D2O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL85365.068.23 / METC23-050
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia; Skeletal Muscle Atrophy; Protein Malnutrition
Keywords: Muscle protein synthesis
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Kwashiorkor | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel-group trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Protein supplements are packed the same and look and taste similar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maltodextrin (Placebo Comparator): daily 2 x 20g maltodextrin ingestion
  Interventions: Behavioral: Resistance exercise; Behavioral: Standardized diet; Dietary Supplement: Maltodextrin supplement
- Milk protein (Experimental): daily 2 x 20g milk protein ingestion
  Interventions: Behavioral: Resistance exercise; Behavioral: Standardized diet; Dietary Supplement: Milk protein supplement
- Plant protein blend (Experimental): daily 2 x 20g plant protein blend ingestion
  Interventions: Behavioral: Resistance exercise; Behavioral: Standardized diet; Dietary Supplement: Plant protein supplement

INTERVENTIONS:
Behavioral: Resistance exercise — 4 single-leg exercise sessions
  Other Names: Strength exercise; Resistance training
Behavioral: Standardized diet — Fully standardized provided energy-balanced diet providing recommended daily allowance for protein.
Dietary Supplement: Plant protein supplement — Dissolved in water with breakfast and prior to sleep.
  Arms: Plant protein blend
Dietary Supplement: Maltodextrin supplement — Dissolved in water with breakfast and prior to sleep.
  Arms: Maltodextrin
Dietary Supplement: Milk protein supplement — Dissolved in water with breakfast and prior to sleep.
  Arms: Milk protein

SUMMARY:
Background Protein intake is important for skeletal muscle mass maintenance with aging and the ingestion of specifically-timed protein supplements could increase overall protein intake and thereby contribute to skeletal muscle mass maintenance. Recently, more attention has been given to the ingestion of plant-based protein blends as a more sustainable high-quality alternative to milk protein, as a means to increase muscle protein build-up and, as such, support muscle maintenance, especially when consuming suboptimal amounts of protein in the regular diet.

Objective To assess the benefit of daily protein supplementation with either a plant-based protein blend or a milk protein on top of a standard diet to stimulate integrated muscle protein synthesis rates in healthy older individuals with and without exercise.

Hypotheses It is hypothesized that both the plant protein blend and the milk protein supplement will result in greater muscle protein build-up when compared with a standard diet control condition.

It is also hypothesized that exercise will result in greater muscle protein build-up when compared to the resting leg in all conditions, with similar effects of the protein supplements vs the control diet as in the non-exercised leg.

This study will show the potential benefit of protein supplementation with alternative protein sources to support skeletal muscle maintenance in older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex
* Aged between 60 and 80 y inclusive
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Following a self-reported vegetarian and vegan diet the 6 months prior to the study.
* Intolerant to milk products
* Corn allergy
* Pea allergy
* Participating currently or in the 3 months prior to the study in a structured (progressive) exercise program.
* Smoking regularly (i.e. >5 cigarettes/week)
* History of cardiovascular, respiratory, gastrointestinal, urogenital, neurological, psychiatric, dermatologic, musculoskeletal, metabolic, endocrine, haematological, immunologic disorders, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol, interfere with the execution of the experiment, or potential influence the study outcomes (to be decided by the principal investigator and responsible physician)
* Diagnosed with phenylketonuria (PKU)
* Uncontrolled hypertension (blood pressure above 160/100 mmHg)
* Donated blood 3 months prior to test day
* Use of any medications that interferes with study participation and/or outcomes (i.e. corticosteroids, non-steroidal anti-inflammatories, gastric acid suppressing medication) as assessed by the responsible medical doctor.
* Use of DOAC, vitamin-K-antagonist, or multiple anticoagulants
* Pregnancy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Integrated muscle protein synthesis rates in the non-exercised leg. | 10 days
  Calculated by the changein deuterium labelled alanine in skeletal muscle protein

SECONDARY OUTCOMES:
Integrated muscle protein synthesis rates in the exercised leg. | 10 days
  Calculated by the change in deuterium labelled alanine in skeletal muscle protein
Dietary protein intake | 10 days
  Assessed by calculating the actual intakes from the provided diet
Dietary fat intake | 10 days
  Assessed by calculating the actual intakes from the provided diet
Dietary carbohydrate intake | 10 days
  Assessed by calculating the actual intakes from the provided diet
Step count | 10 days
  Assessed using a accelerometer
Muscle Crosssectional are | 10 days
  Assessed using Ultrasound

OTHER OUTCOMES:
Age (year) | At baseline
  Interview question
Body mass (kg) | At baseline
  Assessed using scale
Height (m) | At baseline
  Assessed using stadiometer
Body fat % | At baseline
  Assessed using Dexa scan
Lean body mass (kg) | At baseline
  Assessed using Dexa scan
Appendicular lean mass (kg) | At baseline
  Assessed using Dexa scan
Sex | At baseline
  Biological sex checked using interview
Systolic and diastolic blood pressure | At baseline
  Automated measurement

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No